CLINICAL TRIAL: NCT00011518
Title: Bladder Cancer Case Control Study of Arsenic in Water
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 7459-CP-001
Record Dates: First submitted 2001-02-22; First posted 2001-02-26 (Estimated); Last update posted 2006-03-23 (Estimated); Status verified 2006-03

CONDITIONS: Bladder Cancer
Keywords: Arsenic; Bladder Cancer; Drinking Water
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
This study is examining the relationship between ingested arsenic and bladder cancer in two areas of California where a large percentage of the population was exposed to drinking water containing arsenic at low to moderate levels.

DETAILED DESCRIPTION:
Water supplies in many parts of the world contain naturally occurring arsenic. Previous studies have shown that arsenic at high doses can cause cancer of the bladder. The risk at lower doses is unknown. This study is examining the relationship between ingested arsenic and bladder cancer in central Nevada and Kings County, California, two areas where a large percentage of the population was exposed to drinking water containing arsenic at low to moderate levels. Approximately 200 people with bladder cancer and 400 people without bladder cancer will be included. Subjects are interviewed by telephone about past residences, occupations, diet, drinking water consumption, and other lifestyle factors. Arsenic measurements in well water have been collected from the appropriate state agencies and are being matched with residences and drinking water consumption rates to estimate lifetime arsenic exposures for each subject. People with bladder cancer will then be compared to those without to see if people with cancer were more likely to have lived in areas with arsenic in their drinking water.

ELIGIBILITY:
Cases must meet the following criteria:

* Diagnosed with primary bladder cancer from January 1, 1997 until December 31, 2000.
* Live in the following counties at the time of diagnosis: Churchill, Lyon, Mineral, Storey, Douglas, Carson City, Nevada, and Kings County, California
* Ages 20-85 at the time of diagnosis.

Controls will be matched to cases based on gender and five year age groups.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 1997-10; Study Completion 2001-07

CONTACTS AND LOCATIONS:
Locations (1):
- Allan Smith Research Office, Berkeley, California, United States